CLINICAL TRIAL: NCT00252057
Title: Testing the Re-Engineered Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Brian Jack, PI, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-24858
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Results first posted 2009-04-13 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: All
Keywords: rehospitalization; readmission; adverse events; discharge
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Re-engineered hospital discharge (Experimental): Participants received the "Re-Engineered Hospital Discharge", a set of 11 discrete, mutually reinforcing components provided by a Discharge Advocate and re-enforced by a telephone call 2-4 days after discharge by a clinical pharmacist.
  Interventions: Behavioral: Re-Engineered Hospital Discharge
- Standard hospital discharge (No Intervention): Participants received the routine, standard hospital discharge.

INTERVENTIONS:
Behavioral: Re-Engineered Hospital Discharge — The "Re-engineered Hospital Discharge" (Project RED) intervention provides a set of 11 discrete, mutually reinforcing components provided by a Discharge Advocate and re-enforced by a telephone call after discharge by a clinical pharmacist.
  Other Names: RED
  Arms: Re-engineered hospital discharge

SUMMARY:
The purpose of this study is to determine if the "Re-Engineered Discharge" will decrease rehospitalization rates and adverse events of patients leaving Boston Medical Center.

DETAILED DESCRIPTION:
This project responds to the problems of non-standardized care and discontinuity at hospital discharge. Post-discharge adverse events are common and have been well documented. However, to date, there are no studies demonstrating the effectiveness of any procedures or tools designed to reduce them. This work builds on our "Safe Practices Implementation Challenge Grant" in which we developed the "Reengineered Hospital Discharge" tool, a set of 10 discrete, mutually reinforcing components. Hypotheses: The newly designed "Re-engineered Hospital Discharge" intervention will (1) reduce the percentage of patients experiencing a post-discharge adverse event, and (2) reduce subsequent hospital utilization (emergency department visits and rehospitalization) within 30 days following hospital discharge. Population Studied: Patients from a network of Community Health Centers discharged from a general medical service at an urban hospital. The subjects studied represent a low-income, ethnically diverse urban population. This study meets AHRQ guidelines for the inclusion of priority populations in research. Methods: 432 adult patients admitted to the general medical service of Boston Medical Center will be enrolled and randomized to (1) those receiving routine discharge as defined by our "Process Map" (Control Group); and (2) those receiving our "Re-engineered Hospital Discharge" intervention, a set of 10 discrete, mutually reinforcing components provided by a Discharge Advocate and re-enforced by a telephone call 2-4 days after discharge by a clinical pharmacist (Intervention Group). Outcome Measures: The primary patient centered outcomes are: the combined 30-day subsequent hospital utilization (readmission and emergency department use), and health status as measured by the SF-12. Process outcomes include the number and severity of the adverse events related to the discharge 30 days after discharge. Although not a primary outcome, an economic analysis will be completed. Expected Results: This project will provide valuable information about whether the "Re-Engineered Discharge" will reduce adverse events related to discharge and decrease subsequent hospital utilization. Deliverables/Dissemination: An advisory committee of senior Boston Medical Center leaders will oversee the project and, if proven effective, will implement the intervention throughout our Academic Medical Center. The "Re-engineered Hospital Discharge" tool will be widely generalizable and widely disseminated.

ELIGIBILITY:
Inclusion Criteria:

The Project Director will meet with the subject to determine if the patient meets inclusion or exclusion criteria.

Inclusion criteria include are patients who:

1. are over 18 years old;
2. are to be discharged to a community, non-institutionalized setting;
3. report that they desire to be hospitalized in the future if there is a clinical need; and
4. are admitted to Firm B of the BMC Inpatient Service.

Exclusion Criteria:

1. admitted to non-general Medical services at BMC (e.g., orthopedic surgery, obstetrics and gynecology, otolaryngology, general surgery, or psychiatry);
2. requiring hospice, nursing home or other institutional settings upon discharge,
3. who die during the admission,
4. subjects who speak languages other than English;
5. those who indicate that they have no access to a telephone or unable to give a contact telephone number; and
6. those not competent to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jack, MD, Principal Investigator — Boston Medical Center - Family Medicine
Locations (1):
- Boston Medical center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woz S, Mitchell S, Hesko C, Paasche-Orlow M, Greenwald J, Chetty VK, O'Donnell J, Jack B. Gender as risk factor for 30 days post-discharge hospital utilisation: a secondary data analysis. BMJ Open. 2012 Apr 18;2(2):e000428. doi: 10.1136/bmjopen-2011-000428. Print 2012. PMID 22514241
- [Derived] Mitchell SE, Paasche-Orlow MK, Forsythe SR, Chetty VK, O'Donnell JK, Greenwald JL, Culpepper L, Jack BW. Post-discharge hospital utilization among adult medical inpatients with depressive symptoms. J Hosp Med. 2010 Sep;5(7):378-84. doi: 10.1002/jhm.673. PMID 20577971
- [Derived] Jack BW, Chetty VK, Anthony D, Greenwald JL, Sanchez GM, Johnson AE, Forsythe SR, O'Donnell JK, Paasche-Orlow MK, Manasseh C, Martin S, Culpepper L. A reengineered hospital discharge program to decrease rehospitalization: a randomized trial. Ann Intern Med. 2009 Feb 3;150(3):178-87. doi: 10.7326/0003-4819-150-3-200902030-00007. PMID 19189907
- See also: Agency for Healthcare Research and Quality — http://www.ahrq.gov/
- See also: Boston Medical Center — http://www.bmc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited between January 1, 2006 and October 16, 2007, from the general medical floors at Boston Medical Center.
Pre-assignment Details: The baseline interview was conducted after enrollment and prior to group assignment, but it did not affect this assignment or lead to exclusion from the study for any participant. All participants who gave consent and agreed to be in the study were assigned to a group
Period: Overall Study
Arm/Group | Re-engineered Hospital Discharge | Standard Hospital Discharge
Started | 373 | 376
Completed | 370 | 368
Not Completed | 3 | 8
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Death | 1 | 2
Not completed — Participant previously enrolled | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Re-engineered Hospital Discharge | Standard Hospital Discharge | Total
Number analyzed (Participants) | 373 | 376 | 749
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 312 | 314 | 626
  >=65 years | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (15.1) | 49.6 (15.3) | 49.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 199 | 377
  Male | 195 | 177 | 372
Region of Enrollment [Number; unit: participants]
  United States | 373 | 376 | 749

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Rehospitalizations (Emergency Department Visits Plus Hospital Admissions) in the 30 Days After Discharge.
Description: The total number of rehospitalizations (emergency department visits plus hospital admissions) in the 30 days after discharge, compared across study arms. Participants could have more than one rehospitalization in this period; all rehospitalizations for each were counted, making the unit of measure the rehospitalizations and not the participants.
Time Frame: 30 days after discharge
Measure: Number; unit: Total number of rehospitalizations
Arm/Group | Re-engineered Hospital Discharge | Standard Hospital Discharge
Number analyzed (Participants) | 370 | 368
Total number of rehospitalizations | 116 | 166

ADVERSE EVENTS:
Arm/Group | Re-engineered Hospital Discharge | Standard Hospital Discharge
Serious Adverse Events (participants affected / at risk) | 0/373 | 0/376
Other Adverse Events (participants affected / at risk) | 0/373 | 0/376

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No